CLINICAL TRIAL: NCT06928493
Title: Assessment of Children's Dental Anxiety During the Pandemic: A Randomized Controlled Clinical Trial Utilizing Child Drawing: Hospital (CD:H) Picture Test
Brief Title: Are Pediatric Patients' Dental Anxiety Levels Affected by Covid -19 Clinical Conditions?
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Alev Alaçam, Prof. Dr. Pediatric dentistry, Gazi University
Other Study IDs: GU.Ethics Committee 2022.07/1
Record Dates: First submitted 2025-04-14; First posted 2025-04-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Anxiety, Dental
Keywords: anxiety,child
MeSH Terms: conditions — Anxiety Disorders | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pandemic Clinical Conditions (PCC): The oral examination of PCC group was done in an isolated dental environment with white overalls, an FFP3 mask, and a visor.
  Interventions: Other: oral examination
- Conventional Clinical Conditions (CCC): The oral examination of CCC group was done in normal dental environment with a standard white coat and surgical mask.
  Interventions: Other: oral examination

INTERVENTIONS:
Other: oral examination — The pre-examination behaviors and attitudes of the children included in the study were measured by an independent dentist (Ş.Y.İ) using the Frankl Behavior Rating Scale (FS). Following this, the children were randomly divided into two groups PCC and CCC . The oral examination of PCC group was done in an isolated dental environment with white overalls, an FFP3 mask, and a visor. The oral examination of CCC group was done in normal dental environment with a standard white coat and surgical mask.After that, patients were asked to draw themselves or the pediatric dentist who performed the examination. A child psychiatrist (B.A.S.) and a pediatric dentist (R.D) with an internationally valid "Child Drawing Analysis" training certificate evaluated the children's drawings independently.

SUMMARY:
Changes in the dental office environment during the pandemic may affect the children's dental anxiety.

This double-blind, randomized, controlled clinical study aimed to assess children's dental anxiety focusing on changes in the dental office environment with the Child Drawing: Hospital (CD: H) picture test.The results showed that most children exhibited positive or very positive behavior and were not significantly affected by changes in the dental environment or clinical attire. The evaluations from the psychiatrist and dentist using CD: H were highly consistent.

DETAILED DESCRIPTION:
The study involved 120 children aged 5-7 years. All patients and their parents were informed about the purpose and method of the study before the study and signed informed consent forms.

Children's behaviors and attitudes before the dental exam were assessed using the Frankl behavioral scale. The children were then divided into two groups:The Pandemic Clinical Conditions (PCC) group, who were examined in an isolated dental office with special attire, and the Conventional Clinical Conditions (CCC) group, who were examined in a standard dental office with typical clinical attire. After the exam, the children were asked to draw a picture, which was then evaluated by a pediatric dentist and child psychiatrist using CD: H.

The results showed that most children exhibited positive or very positive behavior and were not significantly affected by changes in the dental environment or clinical attire. The evaluations from the psychiatrist and dentist using CD: H were highly consistent.

In conclusion, the changes in the dental office and clinical attire during the pandemic did not significantly impact children's anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

Healthy children children between 5-7 years old no prior dentistry experience children willing to draw picture

Exclusion Criteria:

Children who had mental or physical disabilities children < 5 years old, previous dentist experience who refused to draw picture

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 healthy patient aged 5-7 years who had no prior dentistry experience and whose parents agree to participate in the study,children willing to draw were included the study
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Children's Dental Anxiety During the Pandemic: A Randomized Controlled Clinical Trial Utilizing Child Drawing: Hospital (CD:H) Picture Test | 3 months
  It is aimed to assess children's dental anxiety focusing on changes in the dental office environment with the Child Drawing: Hospital (CD: H) picture test.

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Bodur, Prof. Dr, Study Chair — Gazi University Faculty of Dentistry
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma A, Jain MB. Pediatric Dentistry during Coronavirus Disease-2019 Pandemic: A Paradigm Shift in Treatment Options. Int J Clin Pediatr Dent. 2020 Jul-Aug;13(4):412-415. doi: 10.5005/jp-journals-10005-1809. PMID 33149416
- [Result] Assathiany R, Salinier C, Bechet S, Dolard C, Kochert F, Bocquet A, Levy C. Face Masks in Young Children During the COVID-19 Pandemic: Parents' and Pediatricians' Point of View. Front Pediatr. 2021 Jun 23;9:676718. doi: 10.3389/fped.2021.676718. eCollection 2021. PMID 34249814
- [Result] Alsaleh MM, Sabbarini JM, Al-Batayneh OB, Khader YS. Changes in Behavior Management and Treatment Modalities in Pediatric Dentistry during COVID-19 Pandemic. Int J Clin Pediatr Dent. 2020;13(Suppl 1):S125-S131. doi: 10.5005/jp-journals-10005-1885. PMID 34434029
- [Result] Clatworthy S, Simon K, Tiedeman ME. Child drawing: hospital--an instrument designed to measure the emotional status of hospitalized school-aged children. J Pediatr Nurs. 1999 Feb;14(1):2-9. doi: 10.1016/S0882-5963(99)80054-2. PMID 10063243
- [Result] Azab MM. Influence of different personal protective equipment on children's anxiety in dental office: a randomized controlled trial. BMC Oral Health. 2022 Sep 22;22(1):421. doi: 10.1186/s12903-022-02442-5. PMID 36138354
- See also: References identified — https://pubmed.ncbi.nlm.nih.gov